CLINICAL TRIAL: NCT06473493
Title: The Safety and Efficacy of Compound Alverine Citrate Soft Capsules in the Treatment of Portal Hypertension in Patients With Liver Cirrhosis: a Multicentre, Single-arm, Exploratory Trial s: a Multicentre, Single-arm, Exploratory Trial
Brief Title: The Safety and Efficacy of Alverine in the Treatment of Cirrhotic Portal Hypertension
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai East Hospital (Other); Daping Hospital, Army Medical Center of PLA (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-PH-ALV-2402
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hypertension, Portal
Keywords: Portal hypertension; Alverine; Pharmacological therapy
MeSH Terms: conditions — Hypertension, Portal | interventions — alverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alverine Group (Experimental): Compound Alverine Citrate Capsules (Lejiansu; specification: each capsule contains 60 mg of Alverine Citrate and 300 mg of Simethicone; manufactured by the French company UCB Pharma), 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks
  Interventions: Drug: Alverine

INTERVENTIONS:
Drug: Alverine — 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks
  Other Names: Compound Alverine Citrate Capsules

SUMMARY:
Study Overall Design: This trial is a prospective, multi-center, single-arm, exploratory clinical study. Subjects who meet the inclusion criteria and do not meet the exclusion criteria will receive Compound Alverine Citrate Capsules (Lejiansu; specification: each capsule contains 60 mg of Alverine Citrate and 300 mg of Simethicone; produced by Laboratoires Mayoly Spindler, France) after signing the informed consent form. The dosage is 180 mg/day (1 capsule orally three times a day) for a treatment period of 24 weeks. Apart from the baseline period, efficacy will be evaluated at the end of the 24-week treatment period. Safety assessments will be conducted throughout the trial. The safety evaluation will be performed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 by the National Cancer Institute.

Study Population: Patients with cirrhotic portal hypertension

Intervention: Compound Alverine Citrate Capsules (Lejiansu; each capsule contains 60 mg of Alverine Citrate and 300 mg of Simethicone; manufactured by the French company UCB Pharma), 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks.

Study Objectives: To evaluate the safety and efficacy of Compound Alverine Citrate Capsules in treating portal hypertension in patients with cirrhosis.

Study Endpoints Primary Endpoints

1. Safety Assessment: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation of treatment (evaluated according to CTCAE version 5.0).
2. Efficacy Assessment: The response rate at 24 weeks of treatment, defined as a reduction in HVPG by ≥ 10% from baseline or a reduction to below 12 mmHg.

Secondary Endpoints

1. HVPG Changes: The absolute value and percentage change in HVPG from baseline after 24 weeks of treatment.
2. Decompensation Events: Incidence of cirrhosis decompensation events during treatment, including esophageal/gastric variceal bleeding and re-bleeding, new or worsening ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, and acute kidney injury/hepatorenal syndrome.
3. 12-Week Response Rate: The treatment response rate at 12 weeks.
4. Mortality and Transplantation: Rates of death, liver transplantation, and liver disease-related mortality during the treatment period.

Exploratory Endpoints

1. Cardiac Function: Changes in cardiac function from baseline after 24 weeks of treatment.
2. Liver and Spleen Stiffness: Changes in liver and spleen stiffness from baseline after 24 weeks of treatment.
3. Esophageal Varices: Status of esophageal varices after 24 weeks of treatment.

Sample Size Calculation: This trial is a single-arm, exploratory clinical study, and plans to enroll 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years (inclusive), regardless of gender.
* Patients diagnosed with cirrhosis through clinical evaluation, laboratory tests, imaging studies, and/or liver biopsy.
* Hepatic venous pressure gradient (HVPG) ≥ 12 mmHg.
* Willingness to participate and sign the informed consent form.

Exclusion Criteria:

* Use of non-selective β-blockers (e.g., carvedilol, propranolol) or alverine, papaverine, and its derivatives (e.g., papaverine hydrochloride, drotaverine hydrochloride) within 4 weeks prior to enrollment.
* Previous transjugular intrahepatic portosystemic shunt (TIPS) or other interventional treatments affecting portal pressure (including splenic embolization, microwave treatment of the spleen).
* Previous liver transplantation.
* Occurrence of overt hepatic encephalopathy or esophageal/gastric variceal bleeding within 2 weeks prior to enrollment; endoscopic treatment of esophageal/gastric varices within 1 week prior to enrollment or planned endoscopic treatment.
* Use of somatostatin and its analogs, vasopressin, terlipressin, dopamine, norepinephrine, and other vasoactive drugs within 1 week prior to enrollment.
* History of alcoholism within 12 weeks prior to enrollment and inability to stop drinking during the study (equivalent ethanol intake ≥ 30 g/day for males, ≥ 20 g/day for females).
* Serum total bilirubin level ≥ 3×ULN (for autoimmune liver disease patients, ≥ 5×ULN), serum sodium level < 125 mmol/L, white blood cell count < 1×10^9/L, platelet count < 50×10^9/L, INR > 1.8, or serum creatinine ≥ 1.2×ULN.
* Presence of thrombosis in the portal venous system (including the portal vein, splenic vein, superior mesenteric vein, etc.) or cavernous transformation of the portal vein; previous portal venous system thrombosis if no definite thrombosis detected in the portal venous system within 2 weeks.
* HBV DNA or HCV RNA above the lower limit of detection; patients undergoing active antiviral treatment for hepatitis C; antiviral treatment for hepatitis B < 24 weeks.
* Uncontrollable active infections (e.g., pulmonary infection, abdominal infection, HIV) within 2 weeks prior to enrollment.
* Uncontrolled hypertension, diabetes, or other severe heart/lung diseases.
* Diagnosis or suspicion of malignant tumors, including liver cancer.
* Known allergy to alverine or papaverine and its derivatives (e.g., papaverine hydrochloride, drotaverine hydrochloride) or simethicone.
* Presence of psychiatric symptoms.
* Pregnant or breastfeeding women, or women who may be pregnant.
* Participation in other drug trials within 4 weeks prior to enrollment.
* Any other reasons deemed by the researchers as unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Safety assessment: the incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment. | 24 weeks
  The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment.
24-week response rate | 24 weeks
  The response rate to treatment, defined as the percentage of patients with a decrease in HVPG of ≥10% from baseline or a decrease to below 12 mmHg after 24 weeks of treatment.

SECONDARY OUTCOMES:
HVPG changes: the absolute value change in HVPG from baseline after 24 weeks of treatment | 24 weeks
  The absolute value change in HVPG from baseline after 24 weeks of treatment
HVPG changes: the percentage change in HVPG from baseline after 24 weeks of treatment | 24 weeks
  The percentage change in HVPG from baseline after 24 weeks of treatment
The incidence of decompensation events | 24 weeks
  Incidence of cirrhosis decompensation events during treatment, including esophageal/gastric variceal bleeding and re-bleeding, new or worsening ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, and acute kidney injury/hepatorenal syndrome.
12-week response rate | 12 weeks
  The treatment response rate at 12 weeks
Mortality rate | 24 weeks
  Rates of death and liver disease-related mortality during the treatment period
Transplantation rate | 24 weeks
  Rates of liver transplantation during the treatment period

OTHER OUTCOMES:
Cardiac function changes | 24 weeks
  Changes in cardiac function (LVEF) from baseline after 24 weeks of treatment
Liver stiffness changes | 24 weeks
  Changes in liver stiffness from baseline after 24 weeks of treatment
Spleen stiffness changes | 24 weeks
  Changes in spleen stiffness from baseline after 24 weeks of treatment
Esophageal varices changes | 24 weeks
  Size of esophageal varices after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, M.D., Principal Investigator — Shanghai Changzheng Hospital